CLINICAL TRIAL: NCT04045795
Title: A Multi-center, Open-label, Phase 1b Study to Assess the Pharmacokinetics, Safety, and Efficacy of Subcutaneous and Intravenous Isatuximab (SAR650984) in Combination With Pomalidomide and Dexamethasone, in Patients With Relapsed/Refractory Multiple Myeloma (RRMM)
Brief Title: Multi-center, Open-label, Phase 1b Study in Patients With Relapsed/Refractory Multiple Myeloma (RRMM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TCD15484; U1111-1211-9525 (Registry Identifier: ICTRP); 2018-001996-19 (EudraCT Number)
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; pomalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (5):
- Dose regimen 1 (Experimental): Isatuximab SC administration dose level 1 once weekly for 4 weeks (Cycle 1) and on Day 1 and Day 15 of each subsequent cycle
  Interventions: Drug: pomalidomide; Drug: dexamethasone; Drug: isatuximab SAR650984 SC
- Dose regimen 2 (Experimental): Isatuximab SC administration dose level 2 once weekly for 4 weeks (Cycle 1) and on Day 1 and Day 15 of each subsequent cycle
  Interventions: Drug: pomalidomide; Drug: dexamethasone; Drug: isatuximab SAR650984 SC
- Dose regimen 3 (Experimental): Isatuximab SC administration dose level 3 using the investigational injector device once weekly for 4 weeks (Cycle 1) and on Day 1 and Day 15 of each subsequent cycle
  Interventions: Drug: pomalidomide; Drug: dexamethasone; Drug: isatuximab SAR650984 SC; Device: Investigational injector device
- Dose regimen 4 (Experimental): Isatuximab IV administration once weekly for 4 weeks (Cycle 1) and on Day 1 and Day 15 of each subsequent cycle
  Interventions: Drug: isatuximab SAR650984 IV; Drug: pomalidomide; Drug: dexamethasone
- Dose regimen 5 (Experimental): Isatuximab IV administration once weekly for 4 weeks (Cycle 1) and on Day 1 and Day 15 of each subsequent cycle
  Interventions: Drug: isatuximab SAR650984 IV; Drug: pomalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: isatuximab SAR650984 IV — Pharmaceutical form: solution
  Route of administration: intravenous
  Other Names: Sarclisa
  Arms: Dose regimen 4; Dose regimen 5
Drug: pomalidomide — Pharmaceutical form: tablet
  Route of administration: oral
  Other Names: Pomalyst®
Drug: dexamethasone — Pharmaceutical form: tablet
  Route of administration: oral
  Other Names: Decadron®
Drug: isatuximab SAR650984 SC — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Arms: Dose regimen 1; Dose regimen 2; Dose regimen 3
Device: Investigational injector device — Subcutaneous administration
  Arms: Dose regimen 3

SUMMARY:
Primary Objectives:

* To evaluate the safety and tolerability of isatuximab administered subcutaneously (SC) versus intravenously (IV)
* To assess the safety and tolerability (including local injection site tolerability) of isatuximab using the (investigational) isatuximab injector device
* To evaluate the pharmacokinetics (PK) of SC and IV isatuximab

Secondary Objectives:

* To estimate absolute bioavailability of SC and IV isatuximab
* To measure receptor occupancy (RO) after isatuximab SC versus IV administration
* To assess efficacy of isatuximab after SC and IV administration
* To assess patient expectations prior to and patient experience and satisfaction after SC administration
* To evaluate potential immunogenicity of SC or IV isatuximab

DETAILED DESCRIPTION:
Total study duration is variable depending on treatment and follow-up periods, including 21 days of screening, and treatment period until disease progression, unacceptable adverse reaction or other reason for discontinuation. End of treatment will be 30 days after last administration of investigational medicinal product, or before further anti-myeloma therapy, whichever comes first; approximately 14 months after first study treatment administration.

ELIGIBILITY:
Inclusion criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
* Participant must be above 18 years of age or country's legal age of majority if the legal age is >18 years old, at the time of signing the informed consent.
* Participant has been previously diagnosed with multiple myeloma (MM) based on standard criteria and currently requires treatment because MM has relapsed following a response, according to International Myeloma Working Group (IMWG) criteria.
* Participant has received at least two previous therapies including lenalidomide and a proteasome inhibitor and has demonstrated disease progression on last therapy or after completion of the last therapy.
* Participants with measurable disease defined as at least one of the following:
* Serum M protein ≥ 0.5 g/dL (≥5 g/L).
* Urine M protein ≥ 200 mg/24 hours.
* Serum free light chain (FLC) assay: Involved FLC assay ≥ 10 mg/dL (≥ 100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65).
* Male or female: Contraceptive use by men or women

Exclusion criteria:

* Malignancy within 3 years prior to enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status score >2.
* Inadequate hematological, liver or renal function.
* Serum calcium (corrected for albumin) level above the upper limit of normal (ULN) range.
* Patients with prior anti-CD38 treatment are excluded if:

  * Refractory to anti-CD38 treatment defined as progression on or within 60 days of the last dose of the anti-CD38 or,
  * Intolerant to the anti-CD38 previously received or,
  * Progression after initial response on anti-CD38 therapy with a washout period inferior to 9 months before the first dose of isatuximab SC or IV.
* Participant did not achieve a minimal response or better to at least one of the previous lines of treatment (ie, primary refractory disease is not eligible).
* Received any investigational drug within 14 days or 5 half-lives of the investigational drug, whichever is longer.
* Prior anti-cancer therapy within 14 days.
* Any >Grade 1 adverse reaction unresolved from previous treatments according to the NCI-CTCAE v5.0. The presence of alopecia or peripheral neuropathy ≤ Grade 2 without pain is allowed.
* Previous allogeneic stem cell transplantation with active Graft Versus Host Disease or being under immunosuppressive therapy in the last 2 months previously to the inclusion in the trial.
* Daily requirement for corticosteroids.
* Known to be HIV+ or to have hepatitis A or uncontrolled or active hepatitis B virus (HBV) infection (patients with positive HBsAg [HBsAg] and/or HBV DNA) or active HCV (HCV) infection (positive HCV RNA and negative anti-HCV).
* Active tuberculosis and severe infections requiring treatment with antibiotic parenteral administration.
* Any clinically significant, uncontrolled medical conditions that, in the Investigator's opinion, would expose excessive risk to the patient or may interfere with compliance or interpretation of the study results.
* History of erythema multiforme or severe hypersensitivity to prior immunomodulatory drugs (IMiDs).
* Hypersensitivity or history of intolerance to immunomodulatory drugs (IMiDs), dexamethasone, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study therapy that are not amenable to premedication with steroids and histamine H2 blockers or would prohibit further treatment with these agents.
* Inability to tolerate thromboprophylaxis.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events (AEs) | Baseline to 30 days after last study treatment administration (up to approximately 14 months after first study treatment administration)
  Number of participants with adverse events
Pharmacokinetic (PK) assessment: Ceoi | Baseline to end of treatment (EOT) after isatuximab SC and to Cycle 10 after IV (28 days per Cycle)
  Concentration observed at the end of infusion (Ceoi)
PK assessment: Cmax | Baseline to EOT after isatuximab SC and to Cycle 10 after IV (28 days per Cycle)
  Maximum concentration observed after the first infusion (Cmax)
PK assessment: tmax | Baseline to EOT after isatuximab SC and to Cycle 10 after IV (28 days per Cycle)
  Time to reach Cmax (tmax)
PK assessment: Clast | Baseline to EOT after isatuximab SC and to Cycle 10 after IV (28 days per Cycle)
  Last concentration observed above the lower limit of quantification after the first infusion (Clast)
PK assessment: tlast | Baseline to EOT after isatuximab SC and to Cycle 10 after IV (28 days per Cycle)
  Time of Clast (tlast)
PK assessment: Ctrough | Baseline to EOT after isatuximab SC and to Cycle 10 after IV (28 days per Cycle)
  Concentration observed just before treatment administration during repeated dosing (Ctrough)
PK assessment: AUClast | Baseline to EOT after isatuximab SC and to Cycle 10 after IV (28 days per Cycle)
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to time of the last concentration observed above the lower limit of quantification (ie, Clast) (AUClast)
PK assessment: AUC0 T | Baseline to EOT after isatuximab SC and to Cycle 10 after IV (28 days per Cycle)
  Area under the plasma concentration versus time curve calculated over the dosing interval T (168h or 336h) (AUC0 T)

SECONDARY OUTCOMES:
Estimation of absolute bioavailability of isatuximab | Day 8
  Absolute bioavailability of isatuximab SC, expressed as a percentage, estimated from AUC0-168h obtained after intravenous (IV) and extravascular (EV) administration
Overall response rate (ORR) | From day -21 to day 60 after last study treatment (up to approximately 14 months after first study treatment administration)
  ORR is the proportion of patients with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) using the IMWG response criteria
Duration of response (DOR) | From day -21 to day 60 after last study treatment (up to approximately 14 months after first study treatment administration)
  Time from the date of the first response to the date of first progressive disease (PD) or death, whichever happens first
Time to response (TTR) | From day -21 to day 60 after last study treatment (up to approximately 14 months after first study treatment administration)
  Time from the date of first study treatment to the first response
Time to progression (TTP) | From day -21 to day 60 after last study treatment (up to approximately 14 months after first study treatment administration)
  Time from date of first study treatment to date of first documentation of progressive disease
Overall survival (OS) | From day -21 to day 60 after last study treatment (up to approximately 14 months after first study treatment administration)
  Time from the date of first study treatment to date of death from any cause
Clinical benefit rate (CBR) | From day -21 to day 60 after last study treatment (up to approximately 14 months after first study treatment administration)
  Proportion of patients with sCR, CR, VGPR, PR or minimal response (MR) according to IMWG criteria
Progression free survival (PFS) | From day -21 to day 60 after last study treatment (up to approximately 14 months after first study treatment administration)
  Time from date of first study treatment to date of first documentation of progressive disease or death
Comparison of patient expectations and satisfaction: Patient Expectations and Satisfaction Questionnaires | Cycles 1 and 2 (28 days per Cycle), and 30 days after last isatuximab administration (up to approximately 14 months after first study treatment administration)
  Comparison of patient expectations and satisfaction will be assessed using Patient Expectations and Satisfaction Questionnaires before and after subcutaneous (SC) administration, where a score of 1 = not satisfied and a score of 5 = extremely satisfied
Immunogenicity: Anti drug antibody levels | Baseline to EOT after isatuximab SC and to Cycle 10 after IV (28 days per Cycle)
  Incidence of patients with anti drug antibodies against isatuximab
Biomarker: Change in CD38 receptor occupancy | At screening and at Day 1 of Cycle 2 (28 days per Cycle) (predose); to be stopped once the isatuximab SC dose has been selected.
  Change in CD38 receptor occupancy from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (14):
- United States (3):
  - ~Banner MD Anderson Cancer Center Site Number : 8400005, Gilbert, Arizona
  - City of Hope Site Number : 8400002, Duarte, California
  - Gabrail Cancer Center Site Number : 8400001, Canton, Ohio
- Australia (4):
  - Investigational Site Number : 0360002, Blacktown, New South Wales
  - Investigational Site Number : 0360001, Wollongong, New South Wales
  - Investigational Site Number : 0360004, Fitzroy, Victoria
  - Investigational Site Number : 0360003, Richmond, Victoria
- Investigational Site Number : 0560001, Leuven, Belgium
- France (2):
  - Investigational Site Number : 2500001, Nantes
  - Investigational Site Number : 2500002, Toulouse
- Japan (2):
  - Investigational Site Number : 3920002, Okayama, Okayama-ken
  - Investigational Site Number : 3920001, Shibuya-ku, Tokyo
- Spain (2):
  - Investigational Site Number : 7240002, Santander, Cantabria
  - Investigational Site Number : 7240001, Badalona, Catalunya [Cataluña]

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TCD15484 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25346&tenant=MT_SNY_9011